CLINICAL TRIAL: NCT03030690
Title: A Clinical Assessment of Class II Glass Carbomer Cement Restorations Compared to Resin Modified Glass Ionomer Cement and Composite Resin Restorations in Primary Molars.
Brief Title: A Clinical Assessment of Glass Carbomer Cement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Sumaya Nouri, BDS, M.Sc, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 070-16
Record Dates: First submitted 2017-01-21; First posted 2017-01-25 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Dental Caries Class II
Keywords: Proximal Dental Caries; Glass Carbomer; Hydroxyapatite Enhanced Glass Ionomer; Primary Teeth
MeSH Terms: interventions — glass carbomer cement; Composite Resins; Filtek Z250

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Glass Carbomer Cement (Experimental): GCP Glass Fill, Glass Carbomer™Tech, Ridderkerk, Netherlands
  Interventions: Other: Glass Carbomer Cement
- Resin Modified Glass Ionomer Cement (Active Comparator): GC Fuji II LC Capsule, GC International, Tokyo, Japan
  Interventions: Other: Resin Modified Glass Ionomer Cement
- Composite Resin (Active Comparator): Filtek Z250, 3M ESPE, St Paul, MN, USA
  Interventions: Other: Composite Resin

INTERVENTIONS:
Other: Glass Carbomer Cement — Restoration of proximal lesions in primary molars using glass carbomer cement
  Other Names: GCP Glass Fill; Hydroxyapatite enhance glass ionomer cement
  Arms: Glass Carbomer Cement
Other: Composite Resin — Restoration of proximal lesions in primary molars using composite resin.
  Other Names: Filtek Z250
  Arms: Composite Resin
Other: Resin Modified Glass Ionomer Cement — Restoration of proximal lesions in primary molars using resin modified glass ionomer cement
  Other Names: GC Fuji II LC Capsule
  Arms: Resin Modified Glass Ionomer Cement

SUMMARY:
This study will evaluate the clinical performance of glass carbomer cement restorations in restoring proximal lesions in primary molars compared to that of resin modified glass ionomer cement and composite resin restorations. Teeth will be randomly assigned to one of the three restoration groups and the restorations will be evaluated clinically and radiographically every six months.

DETAILED DESCRIPTION:
Glass Carbomer is a monomer free; carbomised nano-glass restorative cement developed from traditional glass ionomer cement (GIC) and contains nano-sized powder particles of hydroxyapatite and fluorapatite. These materials claim to have improved mechanical properties and better bonding to dentin, in addition to continues fluoride release.

The study is a randomized controlled clinical trial where teeth will be randomly assigned to one of the three restoration groups.

Following medical and dental history, bilateral bitewing radiographs will be taken for each patient to assess the presence of proximal lesions. Suitable teeth will then be randomly assigned to one of the restoration groups. A single operator using local anesthesia and rubber dam isolation will then prepare standardized Class II cavities and place the designated restorations according to the manufacturer's instructions.

The quality of the 3 types of restorations will be clinically evaluated at baseline and every six months for color match, marginal discoloration, anatomic form, marginal adaptation, and secondary caries using the criteria described by "Cvar and Ryge" (2005). The evaluation will be performed by 2 calibrated examiners.

Following placement of the restorations, bitewing radiographs will be taken to evaluate the restorations and will be repeated every six months for detection of recurrent caries.

ELIGIBILITY:
Inclusion Criteria:

* One proximal lesion in a primary molar.
* Radiographic evidence of caries extending at least into the inner half of the enamel but not the inner half of dentin.
* Proximal contact with adjacent healthy or restored teeth.
* Occlusal contact with opposing healthy or restored teeth.
* No indication for pulp therapy or other restorative treatment.
* A predicted survival until exfoliation of 2 years.

Exclusion Criteria:

* Radiographic evidence of caries extending into the inner half of dentin.
* No proximal contact with adjacent healthy or restored teeth.
* No occlusal contact with opposing healthy or restored teeth.
* Tooth indicated for pulp therapy or other restorative treatment.
* A predicted survival until exfoliation of less than 2 years.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
clinical success rate of glass carbomer cement in restoring proximal lesions in primary molars. | 2 Years
  the clinical success of glass carbomer cement in restoring proximal lesions compared to the success of resin modified glass ionomer cement and composite resin.

CONTACTS AND LOCATIONS:
Overall Officials: Najlaa Alamoudi, MSc, DSc, Study Chair — King Abdulaziz University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen X, Du MQ, Fan MW, Mulder J, Huysmans MC, Frencken JE. Caries-preventive effect of sealants produced with altered glass-ionomer materials, after 2 years. Dent Mater. 2012 May;28(5):554-60. doi: 10.1016/j.dental.2012.01.001. Epub 2012 Jan 31. PMID 22300651
- [Background] Chen X, Du M, Fan M, Mulder J, Huysmans MC, Frencken JE. Effectiveness of two new types of sealants: retention after 2 years. Clin Oral Investig. 2012 Oct;16(5):1443-50. doi: 10.1007/s00784-011-0633-9. Epub 2011 Nov 29. PMID 22124610
- [Background] Cvar JF, Ryge G. Reprint of criteria for the clinical evaluation of dental restorative materials. 1971. Clin Oral Investig. 2005 Dec;9(4):215-32. doi: 10.1007/s00784-005-0018-z. No abstract available. PMID 16315023
- [Background] Gorseta K, Glavina D, Borzabadi-Farahani A, Van Duinen RN, Skrinjaric I, Hill RG, Lynch E. One-year clinical evaluation of a Glass Carbomer fissure sealant, a preliminary study. Eur J Prosthodont Restor Dent. 2014 Jun;22(2):67-71. PMID 25134364
- [Background] Gu YW, Yap AU, Cheang P, Khor KA. Effects of incorporation of HA/ZrO(2) into glass ionomer cement (GIC). Biomaterials. 2005 Mar;26(7):713-20. doi: 10.1016/j.biomaterials.2004.03.019. PMID 15350775
- [Background] Hubel S, Mejare I. Conventional versus resin-modified glass-ionomer cement for Class II restorations in primary molars. A 3-year clinical study. Int J Paediatr Dent. 2003 Jan;13(1):2-8. doi: 10.1046/j.1365-263x.2003.00416.x. PMID 12542617
- [Background] Lucas ME, Arita K, Nishino M. Toughness, bonding and fluoride-release properties of hydroxyapatite-added glass ionomer cement. Biomaterials. 2003 Sep;24(21):3787-94. doi: 10.1016/s0142-9612(03)00260-6. PMID 12818551
- [Background] Lucas ME, Arita K, Nishino M. Strengthening a conventional glass ionomer cement using hydroxyapatite. J Dent Res. 2001;80:711.
- [Background] Moshaverinia A, Ansari S, Moshaverinia M, Roohpour N, Darr JA, Rehman I. Effects of incorporation of hydroxyapatite and fluoroapatite nanobioceramics into conventional glass ionomer cements (GIC). Acta Biomater. 2008 Mar;4(2):432-40. doi: 10.1016/j.actbio.2007.07.011. Epub 2007 Aug 25. PMID 17921077
- See also: The longevity of dental restorations: a systematic review. Report 19, NHS Centre for Reviews and Dissemination — https://www.york.ac.uk/media/crd/crdreport19.pdf